CLINICAL TRIAL: NCT01571856
Title: Efficacy of Use of Zinc in the Treatment of Acute Diarrhea in Infants Under Six Months.
Brief Title: Efficacy of Use of Zinc in the Treatment of Acute Diarrhea in Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Pediatrico Albina de Patino (Other)
Responsible Party: Principal Investigator, Giuseppe Grandy, Medical Chief of Nutrition Center, Centro Pediatrico Albina de Patino
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: protzinc2012
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Acute Diarrhea; Acute Gastroenteritis
Keywords: Acute Diarrhea; Zinc; Children
MeSH Terms: interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- zinc sulfate (Active Comparator): zinc sulphate solution.
  Interventions: Drug: Zinc Sulfate
- cornstarch solution (Placebo Comparator): cornstarch powder diluted in distilled water
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Zinc Sulfate — zinc sulfate solution, contains 20 mg. per 5 mL. dosage 2.5 mL. per day.
  Other Names: Suplizinc
  Arms: zinc sulfate
Other: placebo — cornstarch powder diluted in distilled water, dosage 2.5 ml per day
  Arms: cornstarch solution

SUMMARY:
The purpose of this study is to determine the effect of zinc in acute watery diarrhea in children. The investigators will evaluate the effect of product versus placebo.

DETAILED DESCRIPTION:
Background: Acute Gastroenteritis is one of the most and frequent disease in the childhood, today exist strong evidence of beneficial effect of use of zinc in acute diarrhea in children over 6 months. but there are not enough clinical trials to show this beneficial effect on children under 6 months.

Objectives: To evaluate the effect of zinc in the treatment of children under 6 months age with acute diarrhea.

Methods: A randomized clinical trial, controlled, double-blind. The investigators will have two groups of patients : One group will receive zinc plus oral rehydration and the other one will receive placebo plus oral rehydration; the parameters of evaluation are going to be the duration of diarrheal episode, number of diarrhea stools by day, weight of stool, nutritional state.

ELIGIBILITY:
Inclusion Criteria:

* all acute diarrhea

Exclusion Criteria:

* Severe malnourishment
* Severe dehydration
* Systemic infections
* coinfections

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
duration of diarrheal episode | five days
  duration of diarreal episode, time in wich the watery stools will be normalized, an expected average of 5 days.

SECONDARY OUTCOMES:
duration of hospitalization | 5 days
  participants will be followed for the duration of hospital stay, an expected average of 5 days
weight of stool | 5 days
  we expected the weight of the stool will diminish by about 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Grandy, MD MSc, Study Director — Centro Pediatrico Albina de Patino; Zaida Cama, MD, Study Chair — Centro Pediatrico Albina Ptino
Locations (1):
- Centro Pediatrico Albina Patino, Cochabamba, Departamento de Cochabamba, Bolivia